CLINICAL TRIAL: NCT05966298
Title: Investigation of The Efficacy of Core Stabilization Training in Patients With Subacromial Impingement Syndrome: A Randomized Controlled Study
Brief Title: Investigation of the Effectiveness of Core Stabilization Training in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Eren Ozen, Principal Investigator, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-29
Record Dates: First submitted 2023-07-13; First posted 2023-07-28 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial Impingement Syndrome; core stabilization training; core stability; pain; range of motion; upper extremity function; Subacromial Impingement; Impingement; Core Stabilization Exercises; core stability exercises
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Core stabilization group (Experimental): Individuals included in this group will receive 20 minutes of core stabilization training in addition to 40 minutes of standard rehabilitation. Patients will be trained 5 days a week for first 3 weeks(standart rehabilitation + core stabilization training) then will be trained 3 days a week on 4-6 week (only core stabilization training). The next 6 weeks will be given a home exercise program including shoulder exercises and core stabilization training.
  Interventions: Other: Core stabilization training; Other: Standart Rehabilitation
- Control group (Other): Individuals included in this group will receive only 40 minutes of standard rehabilitation. Patients will be trained 5 days a week for first 3 weeks(only standart rehabilitation). The next 9 weeks will be given a home exercise program including shoulder exercises.
  Interventions: Other: Standart Rehabilitation

INTERVENTIONS:
Other: Core stabilization training — First, while focusing on the activation methods of deep cervical flexor, transversus abdominus and multifidus muscles in individuals; In the next stages, exercises will be performed that will preserve the contraction of the deep cervical flexor, transversus abdominus and multifidus muscles and activate the other muscles of the body.
  Arms: Core stabilization group
Other: Standart Rehabilitation — This treatment includes shoulder exercises and conventional therapy (Infrared, TENS).

SUMMARY:
Subacromial Impingement Syndrome (SIS) is one of the most common shoulder problems. The core region is considered a kinetic link that facilitates the transfer of torque and angular momentum between the upper and lower extremities during body movements. The decrease in core stabilization affects both trunk control and the quality of extremity movements depending on the kinetic chain in the body. The improvement in core stabilization balances the load transfer between the trunk and the extremities and reduces the asymmetry between the extremities. Core stabilization training should be included in rehabilitation programs as core stabilization is adversely affected in patients with SIS. For this reason, this study was planned to examine the effects of core stabilization training applied in addition to conventional treatment in patients with SIS on pain, range of motion, shoulder muscles strenght and core stability.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with subacromial impingement syndrome,
* Being between the ages of 18-65,
* Not having received medical treatment,
* Not having received a shoulder-related physiotherapy program in the last 1 year,
* Not having undergone any shoulder-related surgery,
* Being able to read and understand Turkish

Exclusion Criteria:

* Neurological deficits of the upper extremity and the presence of another orthopedic disease, rheumatic and congenital disease other than CNS
* Presence of mental problems,
* To have received corticosteroid treatment in the last year,
* Having cardiovascular and systemic diseases that prevent work,
* Pregnancy,
* Those with communication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline
  It is used to assess the severity of pain. Pain severity with Visual Analogue Scale,(0-10) higher scores indicate more pain.
Visual Analogue Scale | 3 week
  It is used to assess the severity of pain. Pain severity with Visual Analogue Scale,(0-10)higher scores indicate more pain.
Visual Analogue Scale | 6 week
  It is used to assess the severity of pain. Pain severity with Visual Analogue Scale,(0-10)higher scores indicate more pain.
Visual Analogue Scale | 12 week
  It is used to assess the severity of pain. Pain severity with Visual Analogue Scale,(0-10)higher scores indicate more pain.
Digital dynamometer | Baseline
  It will be used to measure the strength of the shoulder muscles.
Digital dynamometer | 3 week
  It will be used to measure the strength of the shoulder muscles.
Digital dynamometer | 6 week
  It will be used to measure the strength of the shoulder muscles.
Digital dynamometer | 12 week
  It will be used to measure the strength of the shoulder muscles.
QuickDASH | Baseline
  It is a questionnaire that evaluates disorders in all upper extremity functions. The QuickDASH is an abbreviated 11-question subset from the original Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. The questionnaire's answers are scored on a 1-5 points scale that is then transformed to result in a score that ranges from 0 (indicating least disability) to 100 (indicating most disability).
QuickDASH | 3 week
  It is a questionnaire that evaluates disorders in all upper extremity functions. The QuickDASH is an abbreviated 11-question subset from the original Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. The questionnaire's answers are scored on a 1-5 points scale that is then transformed to result in a score that ranges from 0 (indicating least disability) to 100 (indicating most disability).
QuickDASH | 6 week
  It is a questionnaire that evaluates disorders in all upper extremity functions. The QuickDASH is an abbreviated 11-question subset from the original Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. The questionnaire's answers are scored on a 1-5 points scale that is then transformed to result in a score that ranges from 0 (indicating least disability) to 100 (indicating most disability).
QuickDASH | 12 week
  It is a questionnaire that evaluates disorders in all upper extremity functions.The QuickDASH is an abbreviated 11-question subset from the original Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. The questionnaire's answers are scored on a 1-5 points scale that is then transformed to result in a score that ranges from 0 (indicating least disability) to 100 (indicating most disability).
Stabilizer pressure biofeedback device | Baseline
  This device will be used to measure deep cervical flexor muscles endurance.
Stabilizer pressure biofeedback device | 3 week
  This device will be used to measure deep cervical flexor muscles endurance.
Stabilizer pressure biofeedback device | 6 week
  This device will be used to measure deep cervical flexor muscles endurance.
Stabilizer pressure biofeedback device | 12 week
  This device will be used to measure deep cervical flexor muscles endurance.
Modified "Biering-Sorensen" test | Baseline
  Test will be applied to assess the endurance of the core muscles. The subjects are positioned in the prone position. The subjects are asked to extend their upper body straight forward from the edge of the table. How long the patient was able to perform the test was recorded in seconds.
Modified "Biering-Sorensen" test | 3 week
  Test will be applied to assess the endurance of the core muscles. The subjects are positioned in the prone position. The subjects are asked to extend their upper body straight forward from the edge of the table. How long the patient was able to perform the test was recorded in seconds.
Modified "Biering-Sorensen" test | 6 week
  Test will be applied to assess the endurance of the core muscles. The subjects are positioned in the prone position. The subjects are asked to extend their upper body straight forward from the edge of the table. How long the patient was able to perform the test was recorded in seconds.
Modified "Biering-Sorensen" test | 12 week
  Test will be applied to assess the endurance of the core muscles. The subjects are positioned in the prone position. The subjects are asked to extend their upper body straight forward from the edge of the table. How long the patient was able to perform the test was recorded in seconds.
Trunk flexors endurance test | Baseline
  Test will be applied to assess the endurance of the core muscles. Participants will be positioned with trunk flexed to 60º, knees and hips to 90º flexion. The evaluator fixes the feet on the ground by supporting them from the toes. When the 60º trunk flexion is broken, the test will be terminated. How long the patient was able to perform the test was recorded in seconds.
Trunk flexors endurance test | 3 week
  Test will be applied to assess the endurance of the core muscles. Participants will be positioned with trunk flexed to 60º, knees and hips to 90º flexion. The evaluator fixes the feet on the ground by supporting them from the toes. When the 60º trunk flexion is broken, the test will be terminated. How long the patient was able to perform the test was recorded in seconds.
Trunk flexors endurance test | 6 week
  Test will be applied to assess the endurance of the core muscles. Participants will be positioned with trunk flexed to 60º, knees and hips to 90º flexion. The evaluator fixes the feet on the ground by supporting them from the toes. When the 60º trunk flexion is broken, the test will be terminated. How long the patient was able to perform the test was recorded in seconds.
Trunk flexors endurance test | 12 week
  Test will be applied to assess the endurance of the core muscles. Participants will be positioned with trunk flexed to 60º, knees and hips to 90º flexion. The evaluator fixes the feet on the ground by supporting them from the toes. When the 60º trunk flexion is broken, the test will be terminated. How long the patient was able to perform the test was recorded in seconds.
Lateral bridge test | Baseline
  Test will be applied to assess the endurance of the core muscles. The subjects were asked to lie on their side, raise their bodies on their forearms and toes and maintain this position(both sides). How long the patient was able to perform the test was recorded in seconds.
Lateral bridge test | 3 week
  Test will be applied to assess the endurance of the core muscles. The subjects were asked to lie on their side, raise their bodies on their forearms and toes and maintain this position(both sides). How long the patient was able to perform the test was recorded in seconds.
Lateral bridge test | 6 week
  Test will be applied to assess the endurance of the core muscles. The subjects were asked to lie on their side, raise their bodies on their forearms and toes and maintain this position(both sides). How long the patient was able to perform the test was recorded in seconds.
Lateral bridge test | 12 week
  Test will be applied to assess the endurance of the core muscles. The subjects were asked to lie on their side, raise their bodies on their forearms and toes and maintain this position(both sides). How long the patient was able to perform the test was recorded in seconds.
Prone bridge test | Baseline
  Test will be applied to assess the endurance of the core muscles. The subjects put their elbows on the ground as the starting position and open their feet about the width of their hips while keeping their body straight. The tests end when the subjects break the test positions. How long the patient was able to perform the test was recorded in seconds.
Prone bridge test | 3 week
  Test will be applied to assess the endurance of the core muscles. The subjects put their elbows on the ground as the starting position and open their feet about the width of their hips while keeping their body straight. The tests end when the subjects break the test positions. How long the patient was able to perform the test was recorded in seconds.
Prone bridge test | 6 week
  Test will be applied to assess the endurance of the core muscles. The subjects put their elbows on the ground as the starting position and open their feet about the width of their hips while keeping their body straight. The tests end when the subjects break the test positions. How long the patient was able to perform the test was recorded in seconds.
Prone bridge test | 12 week
  Test will be applied to assess the endurance of the core muscles. The subjects put their elbows on the ground as the starting position and open their feet about the width of their hips while keeping their body straight. The tests end when the subjects break the test positions. How long the patient was able to perform the test was recorded in seconds.
Modified "Push-ups" test | Baseline
  Test will be applied to assess the strength of the core muscles. The subjects are positioned in the prone position with their hands shoulder-width apart and elbows and knees flexed. The subjects were asked to raise their body up by extending their elbows. The number of times the patient repeats the movement in 30 seconds is recorded.
Modified "Push-ups" test | 3 week
  Test will be applied to assess the strength of the core muscles. The subjects are positioned in the prone position with their hands shoulder-width apart and elbows and knees flexed. The subjects were asked to raise their body up by extending their elbows. The number of times the patient repeats the movement in 30 seconds is recorded.
Modified "Push-ups" test | 6 week
  Test will be applied to assess the strength of the core muscles. The subjects are positioned in the prone position with their hands shoulder-width apart and elbows and knees flexed. The subjects were asked to raise their body up by extending their elbows. The number of times the patient repeats the movement in 30 seconds is recorded.
Modified "Push-ups" test | 12 week
  Test will be applied to assess the strength of the core muscles. The subjects are positioned in the prone position with their hands shoulder-width apart and elbows and knees flexed. The subjects were asked to raise their body up by extending their elbows. The number of times the patient repeats the movement in 30 seconds is recorded.
Sit-ups test | Baseline
  Test will be applied to assess the strength of the core muscles. The subjects are asked to flex the trunk while the knees are flexed in the supine position. During the test, the feet of subjects are stabilized. The number of times the patient repeats the movement in 30 seconds is recorded.
Sit-ups test | 3 week
  Test will be applied to assess the strength of the core muscles. The subjects are asked to flex the trunk while the knees are flexed in the supine position. During the test, the feet of subjects are stabilized. The number of times the patient repeats the movement in 30 seconds is recorded.
Sit-ups test | 6 week
  Test will be applied to assess the strength of the core muscles. The subjects are asked to flex the trunk while the knees are flexed in the supine position. During the test, the feet of subjects are stabilized. The number of times the patient repeats the movement in 30 seconds is recorded.
Sit-ups test | 12 week
  Test will be applied to assess the strength of the core muscles. The subjects are asked to flex the trunk while the knees are flexed in the supine position. During the test, the feet of subjects are stabilized. The number of times the patient repeats the movement in 30 seconds is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Eren Özen, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozen E, Ozen MS, Kaya Mutlu E. The effects of core stabilization training in patients with subacromial impingement syndrome: a single-blind randomized controlled study. Disabil Rehabil. 2026 Feb 10:1-15. doi: 10.1080/09638288.2026.2627617. Online ahead of print. PMID 41667391